CLINICAL TRIAL: NCT03769987
Title: Registry for Advanced Sarcoidosis
Brief Title: Registry for Advanced Sarcodiosis
Acronym: REAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Robert P Baughman, Professor, University of Cincinnati
Other Study IDs: REAS
Record Dates: First submitted 2018-02-01; First posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Sarcoidosis
Keywords: neurosarcoidosis, pulmonary hyeprtension, infliximab, repository corticotropin
MeSH Terms: conditions — Sarcoidosis; Neurosarcoidosis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation — observe patients every 6 months

SUMMARY:
Registry with evaluation and genetic information of patients with advanced sarcoidosis and matched sarcoidosis

ELIGIBILITY:
Inclusion criteria

* Patients with diagnosis of sarcoidosis based on ATS/WASOG criteria 22
* Age ≥ 18 years.
* Life expectancy of at least 2 years.
* Pulmonary function tests (spirometry) within one month of entry or willing to under pulmonary function testing on the day of study enrollment
* Sarcoidosis as characterized as either advanced or non-advanced (see protocol for definition of advanced disease)
* Subjects must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.

Exclusion criteria

* Subjects with a medical disorder, condition, or history of such that would impair the subject's ability to participate or complete this study in the opinion of the investigator
* Inability to comply with the protocol and/or not willing or not available for follow-up assessments.
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Advanced sarcoidosis is defined by the presence of one or more of the following features:
  1. Advanced pulmonary disease as defined by one or more of the following
  2. Symptomatic cardiac disease due to sarcoidosis by either MRI or PET scanning and
  3. Symptomatic neurologic disease
  4. Patients who have received third line therapy (anti-TNF antibodies, rituximab, or RCI)
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Death | 2 years
  Determine how many people die during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Robert Baughman, Study Chair — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No